CLINICAL TRIAL: NCT00563771
Title: Phase IV, Compassionate Use Program of Rasburicase for Treatment of Hyperuricemia in Children and Adolescence Patients With Tumor Lysis Syndrome
Brief Title: Rasburicase for Treatment of Hyperuricemia in Children and Adolescence Patients With Tumor Lysis Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8720
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — rasburicase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rasburicase

SUMMARY:
To provide treatment opportunity to children and adolescent patients with hematologic malignancies by supplying the delayed marketed product and also to observe the efficacy and safety of rasburicase used in the treatment of hyperuricemia

ELIGIBILITY:
Inclusion Criteria:

* Acute hyperuricemia patients before / during chemotherapy for hematologic malignancies ( uric acid greater than 7.5 mg/dL )

  * With a minimum life expectancy of 3 months
  * Having previously signed a written informed consent.

Exclusion Criteria:

* Hypersensitivity to uricase or any of the excipients.
* Known history of G6PD deficiency.
* Previous treatment with Rasburicase or Uricozyme.
* Treatment with any investigational drug within 30 days before planned first Rasburicase administration.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2003-03; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Response will be defined as achievement of normal uric acid levels (less than or = to 7.0mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Choe Seong Choon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Seoul, South Korea